CLINICAL TRIAL: NCT05108493
Title: Efficacy of Dry Needling in the Treatment of Lateral Epicondylitis: A Prospective Randomized Controlled Study
Brief Title: Efficacy of Dry Needling in the Treatment of Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Şeniz Akçay, Study Director, Bozyaka Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/138-11/08/2021
Record Dates: First submitted 2021-10-25; First posted 2021-11-05 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Tennis Elbow; Dry Needling
Keywords: Lateral epicondylitis; Dry needling; Pain
MeSH Terms: conditions — Tennis Elbow; Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling and home exercise (Experimental): The experimental intervention will consist of 3 sessions of dry needling of the lateral epicondyle region, once per week with disposable acupuncture needles (0.25x25mm).
  Range of motion, stretching exercises, ulnar and radial deviation, forearm pronation, supination, elbow extensor, and flexor strengthening exercises will be given to all participants.
  The exercise program will be performed for 10 repetitions 2 times a day. All participants will be advised to continue the exercise program for 12 weeks.
  Interventions: Other: Dry needling; Other: Home exercise program
- Home exercise (Active Comparator): Range of motion, stretching exercises, ulnar and radial deviation, forearm pronation, supination, elbow extensor, and flexor strengthening exercises will be given to all participants.
  The exercise program will be performed for 10 repetitions 2 times a day. All participants will be advised to continue the exercise program for 12 weeks.
  Interventions: Other: Home exercise program

INTERVENTIONS:
Other: Dry needling — Three sessions dry needling of lateral epicondyle region, once per week with disposable acupuncture needles (0.25x25mm).
  Arms: Dry needling and home exercise
Other: Home exercise program — All participants will start the home exercise program during the study period consisting of range of motion exercises for wrist flexion, extension, ulnar and radial deviation, elbow flexion and extensor; forearm supinator, and pronator muscles; stretching exercises. Eccentric strengthening of the wrist flexor extensors, ulnar and radial deviation, forearm pronation, supination, and strengthening exercise training will be given to the elbow extensors and flexors. Progressive strengthening exercises will be added to the program. The exercise program will be terminated with stretching exercises. The exercises will be performed for 10 repetitions 2 times a day, stay in each position for 10 seconds, and rest for 30 seconds between periods. Both groups will be advised to continue the exercise program for 12 weeks.

SUMMARY:
Lateral epicondylitis is painful tendinosis of the main extensor tendon that occurs at the fibro-osseous junction of the outer elbow region. Histopathological samples in patients with chronic lateral epicondylitis show that there is angiofibroblastic degeneration and failure in the normal tendon repair process rather than acute inflammation in this region. It has begun to be accepted that the main factor in lateral epicondylitis is not the inflammatory events but the degenerative process. There are many treatment methods that trigger structural healing in tendinopathies.

In this study, the investigators aimed to evaluate the effect of the dry needling method of the lateral epicondyle region.

DETAILED DESCRIPTION:
Lateral epicondylitis occurs as a result of micro-tears and progressive degeneration caused by repetitive tension, especially at the attachment of the main extensor tendon to the lateral epicondyle. The treatment modality to be used, which causes an increase in functional cells, can prevent the apoptotic process; Thus, it is suggested that there are methods that can reconstruct tendon structure and function. Inflammation can have a positive effect on the healing process in the treatment of lateral epicondylitis. Methods such as prolotherapy and platelet-rich plasma therapy are among the methods that trigger the inflammation process in the lateral epicondyle region and subsequently contribute to the regeneration process. In all these treatments, there is evidence that the local healing process is triggered by the 'needle effect'.

Dry needle therapy is a method that has been widely used in musculoskeletal diseases for many years, and it is one of the safe and cost-effective applications.

In this study, the investigators planned to evaluate the clinical efficiency of dry needling of lateral epicondyle area those are the origin of the extensor muscle groups of the wrist in addition to the home exercise program and to compare the groups in terms of pain severity, functionality, and improvement in handgrip strength with the participants applied for the only home exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Tenderness and pain over lateral epicondylitis and provocation of the lateral elbow pain with one the following tests; resisted middle finger extension, resisted wrist extension, the passive stretch of wrist extensors.
* Participants had a direct radiograph of the elbow within the last 3 months
* Epicondylitis bandage users

Exclusion Criteria:

* History of injection for lateral epicondylitis in the last 6 months
* Radial nerve compression
* History of arm/forearm fracture
* Pregnancy/lactation
* Thrombocytopenia
* Coagulopathy
* Bleeding diathesis
* Neuropathy
* Use of anticoagulants
* Widespread pain syndrome
* History of inflammatory arthritis
* Presence of trauma to the elbow region in the last 3 months
* Statement of the participant that he/she will not be able to continue the follow-ups for the research
* Fear of injection
* Untreated psychiatric illness
* Presence of drug/substance abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
The Patient-Rated Tennis Elbow Evaluation (PRTEE) | 0. week (baseline); 4. week; 12. week
  Change in the Patient-Rated Tennis Elbow Evaluation (PRTEE) questionnaire. PRTEE is a 15-item questionnaire designed to measure forearm pain and disability in patients with lateral epicondylitis. PRTEE allows patients to rate their levels of elbow pain and disability from 0 to 10. The test consists of 2 subscales: 1) Pain subscale [5 items] (0 = no pain, 10 = worst imaginable) 2) Function subscale [Specific activities - 6 items, Usual activities - 4 items] (0 = no difficulty, 10 = unable to do). A total score can be computed on a scale of 100 (0 = no disability).
Visual Analogue Scale | 0. week (baseline); 4. week; 12. week
  Change in the Visual Analogue Scale. Pain on the lateral epicondyle at rest during the day was evaluated with the visual analog scale (VAS 0-10 cm).

SECONDARY OUTCOMES:
Pain free handgrip strength | 0. week (baseline); 4. week; 12. week
  Change in the pain-free handgrip strength. JAMAR hand dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Fikriye Elif Saka, Study Chair — University of Health Sciences Izmir Bozyaka Training and Research Hospital; Kamil Yamak, Study Chair — University of Health Sciences Izmir Bozyaka Training and Research Hospital
Locations (1):
- University of Health Sciences Izmir Bozyaka Training and Research Hospital, Izmir, Karabaglar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jobe FW, Ciccotti MG. Lateral and Medial Epicondylitis of the Elbow. J Am Acad Orthop Surg. 1994 Jan;2(1):1-8. doi: 10.5435/00124635-199401000-00001. PMID 10708988
- [Background] Krogh TP, Bartels EM, Ellingsen T, Stengaard-Pedersen K, Buchbinder R, Fredberg U, Bliddal H, Christensen R. Comparative effectiveness of injection therapies in lateral epicondylitis: a systematic review and network meta-analysis of randomized controlled trials. Am J Sports Med. 2013 Jun;41(6):1435-46. doi: 10.1177/0363546512458237. Epub 2012 Sep 12. PMID 22972856
- [Background] Carayannopoulos A, Borg-Stein J, Sokolof J, Meleger A, Rosenberg D. Prolotherapy versus corticosteroid injections for the treatment of lateral epicondylosis: a randomized controlled trial. PM R. 2011 Aug;3(8):706-15. doi: 10.1016/j.pmrj.2011.05.011. PMID 21871414
- [Background] Navarro-Santana MJ, Sanchez-Infante J, Gomez-Chiguano GF, Cleland JA, Lopez-de-Uralde-Villanueva I, Fernandez-de-Las-Penas C, Plaza-Manzano G. Effects of trigger point dry needling on lateral epicondylalgia of musculoskeletal origin: a systematic review and meta-analysis. Clin Rehabil. 2020 Nov;34(11):1327-1340. doi: 10.1177/0269215520937468. Epub 2020 Jun 23. PMID 32576044
- [Background] Uygur E, Aktas B, Ozkut A, Erinc S, Yilmazoglu EG. Dry needling in lateral epicondylitis: a prospective controlled study. Int Orthop. 2017 Nov;41(11):2321-2325. doi: 10.1007/s00264-017-3604-1. Epub 2017 Aug 21. PMID 28828509
- [Background] Uygur E, Aktas B, Yilmazoglu EG. The use of dry needling vs. corticosteroid injection to treat lateral epicondylitis: a prospective, randomized, controlled study. J Shoulder Elbow Surg. 2021 Jan;30(1):134-139. doi: 10.1016/j.jse.2020.08.044. Epub 2020 Sep 17. PMID 32950674
- [Background] Stoychev V, Finestone AS, Kalichman L. Dry Needling as a Treatment Modality for Tendinopathy: a Narrative Review. Curr Rev Musculoskelet Med. 2020 Feb;13(1):133-140. doi: 10.1007/s12178-020-09608-0. PMID 31942676